CLINICAL TRIAL: NCT00918528
Title: Effect of Mitomycin C on Urethral Stricture Recurrence After Internal Urethrotomy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Nachum Erlich, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0020-09-HYMC
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Urethral Stricture
Keywords: Urethral stricture; Mitomycin C; Internal Urethrotomy
MeSH Terms: conditions — Urethral Stricture

ARMS (2):
- 1. Internal urethrotomy (Active Comparator)
  Interventions: Procedure: Internal urethrotomy
- 2. Internal urethrotomy + mitomycin C (Experimental)
  Interventions: Procedure: Internal urethrotomy; Drug: Mitomycin C - local injection

INTERVENTIONS:
Procedure: Internal urethrotomy
Drug: Mitomycin C - local injection
  Arms: 2. Internal urethrotomy + mitomycin C

SUMMARY:
The aim of this study is to evaluate the efficacy of local injected mitomycin C at the time of internal urethrotomy in order to prevent the recurrence of urethral strictures.

ELIGIBILITY:
Inclusion Criteria:

* Male urethral stricture suitable for internal urethrotomy
* Stricture length less than 10 mm

Exclusion Criteria:

* Stricture length over 10 mm
* Benign prostate enlargement

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-06

PRIMARY OUTCOMES:
Urethral stricture recurrence | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel